CLINICAL TRIAL: NCT01053611
Title: Changes in a Composite Variability Index (CVI) and Bispectral Index (BIS) in Response to Standardized Pain Stimuli During Propofol Remifentanil Infusion
Brief Title: Composite Variability Index Versus Bispectral Index (BIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: M.M.R.F.Struys, University Medical Center Groningen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009.083
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2009-09

CONDITIONS: Sedation During
Keywords: composite variability index; bispectral index; pain
MeSH Terms: conditions — Pain | interventions — Propofol; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Group 1 BIS value 30 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 0 ng/ml
- Group 2 BIS value 30 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 2 ng/ml
- Group 3 BIS value 30 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 4 ng/ml
- Group 4 BIS valaue 30 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 6 ng/ml
- Group 1 BIS value 50 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 0 ng/ml
- Group 2 BIS value 50 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 2 ng/ml
- Group 3 BIS value 50 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 6 ng/ml
- Group 4 BIS value 50 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 6 ng/ml
- Group 1 BIS value 70 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 0 ng/ml
- Group 2 BIS value 70 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 2 ng/ml
- Group 3 BIS value 70 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 4 ng/ml
- Group 4 BIS value 70 (Active Comparator)
  Interventions: Drug: propofol + remifentanil 6 ng/ml

INTERVENTIONS:
Drug: propofol + remifentanil 0 ng/ml — remifentanil 0 ng/ml
  Arms: Group 1 BIS value 30
Drug: propofol + remifentanil 2 ng/ml
  Arms: Group 2 BIS value 30
Drug: propofol + remifentanil 4 ng/ml
  Arms: Group 3 BIS value 30
Drug: propofol + remifentanil 6 ng/ml
  Arms: Group 4 BIS valaue 30
Drug: propofol + remifentanil 0 ng/ml
  Arms: Group 1 BIS value 50
Drug: propofol + remifentanil 2 ng/ml
  Arms: Group 2 BIS value 50
Drug: propofol + remifentanil 6 ng/ml
  Arms: Group 3 BIS value 50
Drug: propofol + remifentanil 6 ng/ml
  Arms: Group 4 BIS value 50
Drug: propofol + remifentanil 0 ng/ml
  Arms: Group 1 BIS value 70
Drug: propofol + remifentanil 2 ng/ml
  Arms: Group 2 BIS value 70
Drug: propofol + remifentanil 4 ng/ml
  Arms: Group 3 BIS value 70
Drug: propofol + remifentanil 6 ng/ml
  Arms: Group 4 BIS value 70

SUMMARY:
The aim of this study is to compare the accuracy of the changes in CVI in response to a standardized noxious stimulus during various targeted pseudo-steady-state concentrations of remifentanil and various steady state level of BIS as guided by propofol effect compartment controlled TCI (closed-loop).

DETAILED DESCRIPTION:
Patients will be allocated to receive a specific effect-site concentration of remifentanil and propofol. For remifentanil, concentrations will be targeted at 0, 2, 4 and 6 ng/ml. After an equilibration period, anesthesia will be induced in all patients using propofol in order to reach and maintain a BIS value of 70, 50 or 30. After an equilibration period(from start of propofol infusion), OAA/S will be measured in all patient. All patients will receive a standard pain stimulus (30 seconds, 50 mA) in order to observe the influence of the effect-site concentration of propofol and remifentanil on the CVI. A time window of 5 minutes after the stimulus will be respected to observe the changes in both BIS and CVI. After this period, the study will be terminated and classical maintenance of anesthesia will be provided.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I and II patients requiring general anesthesia for elective surgical procedures

Exclusion Criteria:

* patient refusal
* weight less than 70% or more than 130% of ideal body weight,
* neurological disorder
* recent use of psycho-active medication, including alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
BIS and CVI. | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Sahinovic MM, Eleveld DJ, Kalmar AF, Heeremans EH, De Smet T, Seshagiri CV, Absalom AR, Vereecke HEM, Struys MMRF. Accuracy of the composite variability index as a measure of the balance between nociception and antinociception during anesthesia. Anesth Analg. 2014 Aug;119(2):288-301. doi: 10.1213/ANE.0000000000000274. PMID 24892803